CLINICAL TRIAL: NCT06325410
Title: Prognostic Factors Influencing the Recurrence Rate and Survival of Patients With Colorectal Cancer: a Single Institution Experience
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, Principal Investigator, Zagazig University
Other Study IDs: #11279-20-11-2023
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal; cancer; recurrence; prognosis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: resection of colorectal cancer — resection of bowel segment and re-anastmosis or stoma formation

SUMMARY:
over the past decade colon cancer has emerged as the second most deadly and the third most common type of cancer in the world with increasing incidence in Egypt due to life style and diet change. some research showed relation between colon cancer recurrence and advanced tumor staging. To investigators knowledge, this is the first time to be done in Zagazig University.

Data was collected from records in a retrospective cohort study

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with newly diagnosed colorectal cancer
* Age > 18 years old
* recurrent cases of colorectal cancer

Exclusion Criteria:

* Pediartric patient less than 18 yr
* In operable or metastatic cancer colon
* No other malignancies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient with newely diagnosed colorectal cancer were followed up after surgery to detect if there was a recurrence prospectively, while patients with recurrent colorectal cancer were studied retrospectively to find out factors influencing the recurrence
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
age | through study completion, an average of 5 years
  age of patients was obtained from medical records
sex | through study completion, an average of 5 years
  sex of patients was obtained from medical records
medical disease | through study completion, an average of 5 years
  co-existing medical disease was obtained from medical records
previous surgery | through study completion, an average of 5 years
  previous surgical history was obtained from medical records
CEA | through study completion, an average of 5 years
  value of carcino-embryonic antigen was recorded
tumor grade | through study completion, an average of 5 years
  tumor grade after resection from pathology report recorded
tumor site | through study completion, an average of 5 years
  tumor site recorded from operative findings
tumor size | through study completion, an average of 5 years
  tumor size was measured by length x width in cm from records
surgical margins of resected tumor | through study completion, an average of 5 years
  safety margins were assessed from pathological examination under microscopy and recorded in pathology reports, it can be free surgical margins ( no tumor cells) or positive surgical margins( presence of tumor cells)
neoadjuvant therapy | through study completion, an average of 5 years
  history of neoadjuvant therapy before surgery from records obtained
adjuvant therapy | through study completion, an average of 5 years
  history of adjuvant therapy post operative obtained from records
diet | through study completion, an average of 5 years
  diet and dietary life style from history
occupation | through study completion, an average of 5 years
  occupation of the patient at time of surgery and if it was changed
family history | through study completion, an average of 5 years
  history taking of family history of cancer disease
type of surgery(laparoscopic or open) | through study completion, an average of 5 years
  type of operation was laparoscopic or open surgery obtained from records
soiling by during surgery | through study completion, an average of 5 years
  by history from records if there was soiling of the field by tumor cells
hand sewen or stappled anastmosis | through study completion, an average of 5 years
  if there was bowel re-anastmosis after surgery, it was done using a stappler or hand sewing sutures. this was obtained from operative data in patient records
post operative complications | through study completion, an average of 5 years
  from records; if there were post operative complication like fecal fistula
site of recurrence | through study completion, an average of 5 years
  site of tumor recurrence was detected
type of resected tumor | through study completion, an average of 5 years
  type of tumor was recorded from pathology reports

CONTACTS AND LOCATIONS:
Overall Officials: Reham Zakaria, PhD, Principal Investigator — faculty of medicine Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available on demand by contacting the principle investigator